CLINICAL TRIAL: NCT06299852
Title: Stereotactic Radiation Therapy for HE2-positive Oligometastatic Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TK01
Record Dates: First submitted 2024-02-25; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: HER2-positive Metastatic Breast Cancer; Oligometastatic Disease
Keywords: HER2-positive; Breast cancer; Oligometastatic
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective group: STR + trastuzumab emtansine 24 hours after the STR (Experimental): STR + trastuzumab emtansine. Patients included in the study will will undergo SRT for up to 2 cycles, depending on the location of the irradiated focus, followed by administration of trastuzumab emtansine at a dose of 3.6 mcg/kg once every 3 weeks, up to 4 total cycles. Targeted therapy with trastuzumab emtansine should commence 24 hours after the completion of SRT.
  Interventions: Drug: Trastuzumab emtansine
- Retrospective group: STR + trastuzumab emtansine > 24 hours after the STR (No Intervention): Patients with oligometastatic HER2+ breast cancer who were treated with trastuzumab-emtansine and who had a history of SRT. Retrospectively, using CT and MRI data, the dynamics of the process will be evaluated according to the RECIST 1.1. Based on the data of the medical documentation of patients, the main statistical indicators will be calculated.

INTERVENTIONS:
Drug: Trastuzumab emtansine — SRT for metastatic foci
  Other Names: SRT
  Arms: Prospective group: STR + trastuzumab emtansine 24 hours after the STR

SUMMARY:
This study involves two non-randomized groups of patients: the observation group and the comparison group. The comparison group will retrospectively include data on 29 patients with oligometastatic HER2-positive breast cancer who received treatment with trastuzumab-emtansine and had a history of SRT.

The prospective part of this study aims to include 29 patients with oligometastatic HER2-positive breast cancer. These patients will undergo SRT followed by the administration of trastuzumab emtansine 24 hours after the SRT.

The combined effect of stereotactic radiation therapy on a metastatic lesion followed by anti-HER2 therapy in the 2nd line - trastuzumab emtansine, remains unexplored. This study plans to evaluate the effectiveness of combining systemic therapy and local control methods (SRT) in patients with oligometastatic HER2-positive breast cancer. It will be the first time the efficacy and toxic profile of this new combined treatment method in this patient population will be studied. This basket trial evaluates trastuzumab emtansine for oligo-metastatic breast cancer with the aim of inducing deep responses, long-lasting disease remissions, and potentially cure.

DETAILED DESCRIPTION:
This study involves two non-randomized groups of patients: the observation group and the comparison group.

The comparison group will retrospectively include data on 29 patients with oligometastatic HER2-positive breast cancer who were treated with trastuzumab-emtansine and had a history of SRT. The dynamics of the process will be evaluated retrospectively using CT and MRI data according to RECIST 1.1 criteria. The main statistical indicators will be calculated based on the patients' medical documentation.

The prospective part of this study aims to include 29 patients with oligometastatic HER2-positive breast cancer. These patients will undergo SRT for up to 2 cycles, depending on the location of the irradiated focus, followed by administration of trastuzumab emtansine 3.6 mcg/kg once every 3 weeks, up to 4 total cycles. Trastuzumab emtansine therapy will be initiated 24 hours after the end of the course of SRT. Tumor foci will be assessed according to RECIST 1.1 criteria.

Objective response, general condition, and adverse events will be evaluated before, during, and after treatment.

Patients will be stratified by age, location of metastatic foci, and treatment. Outpatient patient records, medical histories, clinical and laboratory examination data, morphological examination data, CT findings, MRI findings will be used as sources of information for analyzing the results of diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age and able to give written informed consent and comply with study procedures;
2. Clinical diagnosis: breast cancer, metastatic form;
3. Oligo-metastatic disease as determined by standard of care diagnostics, limited to 5 total individual distant metastases, either in one organ or in 2-3 organ systems. Clustered lymph nodes that can be irradiated with curative intent in a single field are defined as single lesion;
4. Possibility of complete elimination of all foci;
5. HER2 expression level of 3+ points according to immunohistochemical analysis (IHC) and/or degree of amplification ≥2.0 according to the results of in situ hybridization (ISH);
6. Patients with stable metastatic brain foci for at least 4-6 weeks (according to MRI);
7. Patients with HER2+ inoperable locally advanced or metastatic breast cancer who previously received taxanes and trastuzumab;
8. ECOG 0-1 status;
9. Life expectancy of more than 6 months.

Exclusion Criteria:

1. T-DM1 therapy in the medical history;
2. Autoimmune diseases in the medical history or treatment of exacerbations during the last three months;
3. Uncontrolled brain metastases and/or carcinomatous meningitis, causing neurological symptoms;
4. Primary multiple malignant tumors: other malignant neoplasms requiring active treatment;
5. Acute myocardial infarction, acute cerebrovascular accident, uncorrectable coagulopathy, decompensated concomitant pathology, infectious diseases in the active phase, ECOG status > 2;
6. Pregnancy, lactation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 month
  Objective response rate is defined as the proportion of participants who have a confirmed CR or PR, as determined by investigator assessment, per RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 month
  Progression free survival (PFS) is defined as the time from the start of study treatment until the disease progression or death.
Toxicity profile | 3 month
  The assessment of adverse events will be carried out according to the STS AE v.5.0 system.
Second co-primary outcome measure is quality of life | 3 month
  of Cancer (EORTC) Quality of Life Questionnaire for Cancer patients with 30 items (QLQ-C30) sum score

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No